CLINICAL TRIAL: NCT05939323
Title: Correlation Study of Family Communication Disorders and Negative Network Use Behavior Among Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 202310892
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Adolescent
Keywords: Adolescents; family communication disorders; negative network use behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Investigation Team: Questionnaires assessed adolescents and their parents ①Adolescents aged 14-25 years old (including 14,25 years old) and their parents, who agreed to participate in the study
  ②Investigate whether they have family communication difficulties and whether they have negative internet use behaviors

SUMMARY:
The entry point of this project is the social background of the post-epidemic era, with teenagers and parents as the research object, aims to explore the relationship between family communication disorders and adolescent negative network use behavior in the post-epidemic era. This project intends to investigate whether there are family communication disorders and negative Internet use behaviors among 14-25 year old teenagers by issuing questionnaires (sample size: 140). In order to conclude whether there is some connection between family communication disorder and adolescent negative network use behavior.

DETAILED DESCRIPTION:
This research project takes the "post-epidemic era" as the background entry point, and explores the relationship between teenagers' negative Internet use behavior and family communication by using questionnaires. Through literature review, it is obtained that family communication disorders may be related to adolescents' emotional changes with their parents, limited peer interaction, and changes in the structure of their lives. In order to avoid the negative feelings brought by family communication barriers, adolescents tend to turn to other areas such as virtual networks to compensate and regain happiness, which can easily lead to negative Internet use behaviors if they are not careful. By studying the "loss of compensation" model proposed by Chinese scholar Gao Wenbin, the application of the "loss of compensation" model to family communication disorders and adolescents' negative Internet use behavior is derived. In this context, if we can study the correlation between family communication barriers and adolescents' negative Internet use behaviors, it will be beneficial to ease the parent-child relationship, correct adolescents' negative Internet use behaviors, and promote the healthy growth of adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14-25 (including 14,25 years old) and their parents;
* Agree to participate in the studies

Exclusion Criteria:

* Persons of interest with a history of prior psychiatric illness, who are suffering from a serious acute illness, are unconscious, emotionally unstable, and unable to communicate normally

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: General adolescents between 14-25 years old and their parents
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Parent-child communication skills | Baseline
  Parent-Child Communication Skills Subscale with 20-item will be used to measure Parent-child communication skills. The scale uses Likert 4 comments, higher dimension scores indicate better communication ability.
Parent-child communication quality | Baseline
  The Parent-Child Communication Quality Subscale with 12 items will be used to measure the communication skills of fathers, mothers and children separately. The scale uses Likert 4 comments, higher dimension scores indicate higher quality of parent-child communication in terms of relationship enhancement or problem solving.
Parent-child communication system subscales | Baseline
  The Parent-Child Communication System Subscale with 18 items will be used to measure the relationship between father-child communication and mother-child communication. The scale uses Likert 4 comments, the larger the difference, the greater the difference in parental roles and the greater the imbalance in communication status.
Social support received by adolescents | Baseline
  The 17-item Adolescent Social Support Scale will be used to measure the support received by adolescents in society. The scale uses 5-point scale, higher scores indicate better social support.
Peer communication | Baseline
  A 24-item Peer Attachment Scale will be used to measure adolescents' communication with their peers. The scale uses 5-point scale, higher scores indicate higher quality of peer attachment.
Internet addiction among adolescents | Baseline
  The 26-item Chinese Internet Addiction Scale will be used to measure the situation of Internet addiction among adolescents. The scale uses Likert 4 comments, higher scores indicate a higher propensity for Internet addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No